CLINICAL TRIAL: NCT05735899
Title: Evaluation of the Safety and Efficacy of Meniscal Preservation Surgery to Correct Meniscal Extrusion
Brief Title: Evaluation of the Safety and Efficacy of Meniscal Preservation Surgery
Status: Recruiting | Type: Observational
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Meniscal Extrusion
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Meniscal Extrusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Core Treatment Group: This is the only group in this study. Participants will receive full standard of care meniscal repair, followed by assessment interventions- ultrasound, MRI, and physical assessment to document healing progress. Participants will return for standard of care post-operative visits with the physician- 6 weeks, 6 months, and 1 year after the operation is performed- at which point the aforementioned interventions will be completed.

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of surgical meniscal preservation techniques to correct meniscal extrusion. The primary endpoint for safety will be analysis of the total number and types of adverse events (AEs) and serious adverse events (SAEs). The primary endpoint for efficacy will include analysis of patient report outcome measures (PROMs).

H0 - Participants undergoing surgical meniscal preservation to correct meniscal extrusion will not exhibit a limited number of safety events nor have favorable outcomes.

H1- Participants undergoing surgical meniscal preservation to correct meniscal extrusion will exhibit a limited number of safety events and have favorable outcomes.

DETAILED DESCRIPTION:
Treatment for meniscal extrusion varies on a patient-by-patient basis as it is generally dependent on the underlying cause of the extrusion. Extrusion should be detected early and treated appropriately. If left untreated irreversible loss of articular cartilage can ensue leading ultimately to osteoarthritis (OA). Meniscal extrusion is not commonly seen in isolation, but rather in association with meniscal tears or OA. Statistically speaking, the most common meniscal pathology associated with extrusion is posterior horn tearing. The goal of surgery with these two diagnoses is to debride and repair the root tear but also to correct the extrusion. Ignoring the extrusion while only fixing the root tear will increases the patient's chances of developing OA in the future. Surgeries repairing larger tears such as radial tears should also look to correct the noted extrusion and restore overall function for long-term patient meniscal health. The primary operative means of treatment for meniscal extrusion relies on centralization of the extruded meniscus. Centralization refers to the restoration of the meniscus to its native position on the tibial plateau. Ozeki et al. looked to accomplish centralization of extruded medial menisci via the pull-out suture technique. Koga et al noted significant positive outcomes in a prospective study on patients undergoing lateral meniscal centralization. This technique involved placing suture anchors on the edge of the tibial plateau with suture loops passing through the meniscocapsular junction. After the anchor knots were placed, the body of the meniscus was then centralized and stabilized in its anatomic position thereby restoring proper meniscal function. Surgical techniques for the treatment of meniscal extrusion continue to advance and represent areas of future investigation.

As previously mentioned, meniscal injury and meniscal extrusion are prevalent amongst middle-aged and elderly people and represent one of the most important risk factors for the development of OA. After failing conservative treatment options, knee replacement is the surgical intervention utilized by orthopaedic surgeons to treat pain and loss of function associated with OA. According to data published by Blue Cross Blue Shield, the average cost associated with an inpatient total knee replacement (TKR) is $30,249. With estimates that 3.5 million TKR surgeries will be performed annually in the United States by 2040, healthcare costs associated with OA are likely to continue to rise without the development of new treatment methods.

Advances in the treatment of previously irreparable meniscal injuries and the identification of meniscal pathology provide potential measures to delay the onset of OA. Reduction in the prevalence of OA will lead to decreased annual spending on healthcare costs associated with OA and TKR. Reduction in the prevalence of OA will also improve productivity in the workforce as well as keeping non workers active in enjoying the many outdoor recreational activities in the state of Florida. Thus, the aim of this study is to evaluate the long-term safety and efficacy of patients undergoing surgical meniscal preservation to correct meniscal extrusion.

ELIGIBILITY:
Inclusion Criteria Patients 18 years or older who are scheduled to have arthroscopic knee surgery to correct meniscal extrusion and preserve the meniscus by one of the investigating physicians will be screened for participation in this study.

Exclusion Criteria

Exclusion criteria will include:

* Participants requiring surgery for either anterior cruciate ligament (ACL) or posterior cruciate ligament (PCL) reconstruction
* Participants with a history of an autoimmune disease
* Participants with a history of diabetes
* Participants with a history of a blood/clotting disorder
* Participants with a history of previous surgery on the injured knee
* Participants with advanced knee OA or excessive knee malalignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Andrews Institute physicians' practices
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS-Pain and Functioning Questionnaire) | 6 weeks post-op timepoint
  PROMIS Pain and Functioning Questionnaire used in this study to to assess overall health functioning and rehabilitation levels of each participant
Patient Reported Outcomes Measurement Information System (PROMIS-Pain and Functioning Questionnaire) | 6 months post-op timepoint
  PROMIS Pain and Functioning Questionnaire used in this study to to assess overall health functioning and rehabilitation levels of each participant
Patient Reported Outcomes Measurement Information System (PROMIS-Pain and Functioning Questionnaire) | 12 months post-op timepoint
  PROMIS Pain and Functioning Questionnaire used in this study to to assess overall health functioning and rehabilitation levels of each participant
Ultrasound | 6 weeks post-op timepoint
  US is a non-invasive and cost-effective imaging modality that allows the physician to assess anatomic structures of the knee such as the meniscus. The meniscotibbital ligament lesion(MTLL) will be measured using ultrasound.
Ultrasound | 6 months post-op timepoint
  US is a non-invasive and cost-effective imaging modality that allows the physician to assess anatomic structures of the knee such as the meniscus. The meniscotibbital ligament lesion(MTLL) will be measured using ultrasound.
Ultrasound | 12 months post-op timepoint
  US is a non-invasive and cost-effective imaging modality that allows the physician to assess anatomic structures of the knee such as the meniscus. The meniscotibbital ligament lesion(MTLL) will be measured using ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrews Institute for Orthopaedics & Sports Medicine, Gulf Breeze, Florida, United States